CLINICAL TRIAL: NCT03228706
Title: Effectiveness of a Structured Group-Based Intervention "Know Your Medicine - Take It For Health" (KYM-TIFH) in Improving Medication Adherence Among Malay Patients With Underlying Type 2 Diabetes Mellitus in the Sarawak State of Malaysia: A Randomized Controlled Trial
Brief Title: Effectiveness of an Intervention in Improving Medication Adherence Among Malay Patients With Underlying Type 2 Diabetes Mellitus in Malaysia
Acronym: MedAdh-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: University Malaysia Sarawak (Other)
Responsible Party: Principal Investigator, Ting Chuo Yew, Principal Assistant Director (Pharmacy Enforcement), Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 35875
Record Dates: First submitted 2017-05-18; First posted 2017-07-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Medication Adherence; Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Medication Adherence; Malay patients; Structured Group-Based Intervention; Randomised controlled trial
MeSH Terms: conditions — Medication Adherence; Diabetes Mellitus, Type 2 | interventions — Health

STUDY DESIGN:
Intervention Model Description: To achieve the objectives, positivist approach with experimental study design will be employed. In specific, it is a double blinded, randomized controlled trial (RCT) which involve two study sites. Nonetheless, the reporting of the SGBI will be in accordance with the checklist recommended by Borek et al. (2015).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A person who is independent of this study and invited by principal investigator will carry out the randomization based on the list of participants who are eligible and agreed to participate. The list of participants with their randomization information will be kept by the committee member without informing any of the researchers including principal investigator or respondents to assure the blinding of both parties throughout the study. On the day of the intervention, that person will register the attendance of respondents and inform them about the actual venue of the program without informing the researchers or the facilitators of the KYM-TIFH. Each HCKS and HCKS will have two venues prepared and available during the period of the study with one venue allocated for intervention group and the other one with for control group. None of the respondents were aware of the difference between the with assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): All the participants who are randomly assigned to the intervention group will be undergoing the Know Your Medicine-Take it for Health (KYM-TIFH) program, which is a one-off structured group-based intervention (SGBI).
  Interventions: Behavioral: Know Your Medicine - Take It For Health (KYM-TIFH)
- Control Group (No Intervention): All the participants who are randomly assigned to the control group will not be given any information related to KYM-TIFH. However, they will be assigned to the venue for the control group and will be asked to fill in questionnaires with the assistance of four facilitators. A briefing on how to answer the questionnaire will be given by the main facilitator and all facilitators are allowed to answer any questions raised by respondents related to the questionnaire. However, they are not allowed to answer on behalf of the respondents. After the completion of the questionnaire, they will be informed about the subsequent follow-up measurement after three, six and twelve months. After that, they will be dismissed and having usual care provided by the health clinic as before without any changes.

INTERVENTIONS:
Behavioral: Know Your Medicine - Take It For Health (KYM-TIFH) — The KYM-TIFH employed psychosocial, educational and behavioral approach. It was designed based on the application of multiple behavior change theories and persuasion theory as recommended by Slater (1999). The cross-theoretical framework for the message design of intervention as recommended by Slater (1999) involved theories such as Transtheoretical Model (TTM) (Prochaska & Velicer 1997), Theory of Reasoned Action (TRA) (Ajzen & Fishbein 1980), Protection Motivation Theory (PMT) (Rogers 1975), Elaboration-Likelihood Model (ELM) (Petty and Cacioppo 1986) and Social Cognitive Theory (SCT) (Bandura 1992) as in Table 2. Nonetheless, the intervention embraces the philosophy of patients' empowerment, which had found to be effective in engaging patients to produce behavioral change among diabetes patients (Anderson 1995; Anderson et al 1995). Hence, the facilitators are trained to employ a non-didactic approach in facilitating the and eliciting the learning among the group members.
  Arms: Intervention Group

SUMMARY:
Poor medication adherence (MA) among Type 2 Diabetes Mellitus (T2DM) patients had found to be gnarly and devastating (Krass et al 2015; Sharma et al 2014). It was estimated that more than half of the patients failed to achieve recommended glycaemic goals due to nonadherence (García-Pérez 2013; World Health Organization 2003). Furthermore, greater adherence rate was significantly associated with better glycemic control, fewer hospital visits and admissions, and lower medical costs. On the other hand, lower adherence rate was significantly associated with poor medication tolerance, the frequency of medication intake (> 2 times a day), having concomitant depression and negative belief about the medications. Consequently, patients who poorly adhere to medications would take more medications due to the poor glycemic control and development of micro- and macrovascular complications (American Diabetes Association 2013). Such condition would further worsen their adherence due to more complex medications and a greater chance of experiencing drug-related side effects (García-Pérez 2013). This inevitably increases the economic burden and wastage to the healthcare system (Meng et al 2017). Hence breaking the vicious cycle is an urgent call to all stakeholders.

Notably, Ministry of Health Malaysia (MOH) had initiated several interventions in curbing the MA problems at national level. One of those which has been perpetuated and led by pharmacists is "Know Your Medicine" (KYM) Campaign since 2007. The national KYM campaign aims to promote the quality use of medicines through mass communication and group-based approach. The messages conveyed include information on their medication management such as why, how and when to take medicines, reporting adverse drug events, awareness on the rational use of medicines and medications that need special precautions. In specific, assuring and improving medication adherence among patients is one of the important components of the campaign (PSD 2008).

In term of improving medication adherence among Malay T2DM patients, a structured group-based intervention (SGBI) called "Know Your Medicine - Take It For Health" with abbreviation KYM-TIGF, was created by the researchers of this study who work at Sarawak Pharmaceutical Services Division in 2016 under the KYM campaign. The KYM-TIGF is a theoretical based, patient empowerment, culturally appropriate and a combination of psychosocial, educational and behavioral intervention. It is a one-off SGBI that aims to improve the medication adherence through the message specially designed with a cross-theoretical framework as recommended by Slater (1999). The model to measure the effectiveness of the SGBI is an integrated model with Theory of Planned Behaviour (Ajzen 1991) as main theory and Information-Motivation-Behavioural Skills Model (Fisher et al. 2006) as supporting theory. The primary outcome of this study is the HbA1c. The secondary outcomes of this study are the medication adherence level as well as the psychosocial variables of the integrated model which include attitude to medication adhere, the subjective norm to medication adherence, perceived behavioral control towards medication adherence, adherence information, adherence skill and intention to adhere.

DETAILED DESCRIPTION:
A current systematic review by Odgers-Jewell et al (2017) revealed that little had been done to investigate the effectiveness of group based education in improving medication adherence among T2DM patients. This concur with the comprehensive review on interventions to improve medication adherence by Conn & Ruppar (2017), as the researchers conclude that there is an urgent need in evaluating the interventions to improve medication adherence that employs group-based approach.

The evidence on the effectiveness of the KYM-TIFH in promoting medication adherence among T2DM patients remain lacking. Furthermore, the current measurement on the effectiveness of the campaign is the increment of the awareness level of public towards proper use of medicines (PSD 2013) without measuring the impact of the campaign on actual behavior change.

Besides aforementioned, Malay ethnic was found to be the main contributor to the prevalence of poor MA (PSD 2013) due to forgetfulness (75.3%) and reluctant to take prescribed medications (43.8%). Facing the high prevalence of poor MA among Malay patients, an effective and efficient approach which could engage more patients within a shorter period of times to improve the medication adherence problems is highly preferred (Odgers-Jewell 2017). Hence, all the problem statements addressed above lead to the necessity of conducting this study, which aims to investigate the effectiveness of the SGBI "KYM-TIFH" in improving MA among Malay patients with T2DM.

Based on the problems stated above, this study aims (1) to measure the effectiveness of MEDIHEALTH in improving the medication adherence level and the component of the extended TPB, (2) to identify the component of the extended TPB that predicts medication adherence after participating in MEDIHEALTH, and (3) to investigate the sustainability of the program.

Based on the first specific objective, ten hypotheses are to be tested:

H1a: Increase in intention to adhere would be mediated by improvements in attitude towards adherence after baseline, which is achieved by participating in MEDIHEALTH.

H1b: Increase in intention to adhere would be mediated by improvements in subjective norm towards adherence after baseline, which is achieved by participating in MEDIHEALTH.

H1c: Increase in medication adherence would be mediated by improvements in intention to adhere after baseline, which is achieved by participating in MEDIHEALTH.

H1d: Increase in intention to adhere would be mediated by improvements in perceived behavioural control towards adherence after baseline, which is achieved by participating in MEDIHEALTH.

H1e: Increase in intention to adhere would be mediated by improvements in adherence information after baseline, which is achieved by participating in MEDIHEALTH.

H1f: Before the intervention, there are no significant differences of medication adherence level and the psychosocial variables related to it among the participants between the intervention group and the control group.

H1g: After 3, 6 and 12 months of the program, the medication adherence levels among the participants in the intervention group are significantly greater than the medication adherence levels before the intervention.

H1h: After 3, 6 and 12 months of the program, the medication adherence levels among the participants in the intervention group are significantly greater than the medication adherence levels of the participants in the control group.

H1i: After 3, 6 and 12 months of the program, the HbA1c levels among the participants in the intervention group are significantly greater than the HbA1c before the intervention.

H1j: After 3, 6 and 12 months of the program, the HbA1c levels among the participants in the intervention group are significantly greater than the HbA1c levels of the participants in the control group.

For the second specific objective, eight hypotheses are to be tested:

H2a: Improvement in attitude towards adherence will contribute to the increase in intention to adhere.

H2b: Improvement in subjective norm towards adherence will contribute to the increase in intention to adhere.

H2c: Improvement in perceived behavioural control towards adherence will contribute to the increase in intention to adhere.

H2d: Improvement in perceived behavioural control towards adherence will contribute to the increase in medication adherence.

H2e: Improvement in intention to adhere will contribute to the increase in medication adherence.

H2f: Improvement in adherence information will contribute to the increase in perceived behavioural control towards adherence.

H2g: Improvement in adherence information will contribute to the increase in medication adherence.

H2i: Improvement in medication adherence level will contribute to the decrease in HbA1c level.

Operational definitions:

1. Medication adherence: Medication adherence is defined as the level of patients in complying with the medications prescribed by healthcare providers. Such level of compliance is measured through 13 items self-efficacy for appropriate medication use scale (Risser et al., 2007) which had been validated among chronic patients with low literacy.
2. T2DM Malay patients: Type 2 Diabetes Mellitus Malay patients of this study refers to all the patients who are prescribed with oral anti-hyperglycaemic agents (OHA) and obtain their medications supply from the pharmacy department of Kota Samarahan Health Clinic (KS-HC) and Petra Jaya Health Clinic (PJ-HC) during the study period. Such T2DM patients whose identity card show their religion as Islam, will be considered as Malay T2DM patients for this study.
3. Structured group based intervention: The structured group based intervention of this study refers to the program "Know Your Medicine - Take it for Health" which was formulated and employed by the Pharmaceutical Services Division of Sarawak State Health Department in late 2016 under the national campaign "Know Your Medicine" to promote medication adherence among T2DM Malay patients. The official name of the intervention is "Kenali Ubat Anda - Ambillah untuk Kesihatan" in Malay language or "Know Your Medicine - Take it for Health" in English with abbreviation KYM-TIFH.
4. Effectiveness: The effectiveness of this study refers to the improvement of HbA1c and medication adherence level among T2DM Malay patients before and after the SGBI with such improvement having a significant difference as compared to the results in control group. Furthermore, the effectiveness of the SGBI will be complemented by the qualitative data through focus group discussion and a semi-structured interview.
5. Complications: The complications in this study refers to the diabetes-related complications including retinopathy, nephropathy, diabetic foot problems, ischemic heart disease and stroke that had been diagnosed by doctors and were documented in patients' medical records during the period of study.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > 7 %
* Malay T2DM patients > 18 years old
* Poor medication adherence (self-efficacy for appropriate medication use scale scoring < 26)

Exclusion Criteria:

* Pregnant Women
* Patients less than 18 years old
* Patients who had severe and enduring mental health problems
* Patients who can't listen or read due to inherited disabilities or malfunction
* Patients who unable to communicate in the Malay language
* Patients who are participating in other studies
* Patients who decline the consent to participate
* Hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c level at baseline, and at 3, 6 and 12 months after intervention. | Measured during the recruitment of participants and after 3, 6 and 12 months of the intervention.
  The HbA1c level before the intervention and after three, six and twelve months of the intervention.
Change of medication adherence at baseline, and at 3, 6 and 12 months after intervention. | Intervention group: measured right before and 3,6 and 12 months after the program. Control group: measured measured right before and 3,6 and 12 months after the program
  The medication adherence is measured by self-efficacy for appropriate medication use scale (Risser et al., 2007).

SECONDARY OUTCOMES:
Change of adherence information at baseline, and at 3, 6 and 12 months after intervention. | Intervention group: measured right before and 3,6 and 12 months after the program. Control group: measured measured right before and 3,6 and 12 months after the program
  The adherence Information is measured using a 6 items 5 points Likert scale adopted from McPherson et al. (2008). It is measured right before the interventional program begin and right after the interventional program finish.
Change of attitude towards medication adherence at baseline, and at 3, 6 and 12 months after intervention. | Intervention group: measured right before and 3,6 and 12 months after the program. Control group: measured measured right before and 3,6 and 12 months after the program
  The attitude towards medication adherence is measured using a 5 items 5 points Likert scale adopted from Farmer et al. (2006). It is measured right before the interventional program begin and right after the interventional program finish.
Change of subjective norms towards medication adherence at baseline, and at 3, 6 and 12 months after intervention. | Intervention group: measured right before and 3,6 and 12 months after the program. Control group: measured measured right before and 3,6 and 12 months after the program
  The subjective norms towards medication adherence is measured using a 6 items 5 points Likert scale adopted from Farmer et al. (2006). It is measured right before the interventional program begin and right after the interventional program finish.
Change of perceived behavioural control towards medication adherence at baseline, and at 3, 6 and 12 months after intervention. | Intervention group: measured right before and 3,6 and 12 months after the program. Control group: measured measured right before and 3,6 and 12 months after the program
  The perceived behavioural control towards medication adherence is measured using a 11 items 5 points Likert scale adopted from Fernandez et al. (2008). It is measured right before the interventional program begin and right after the interventional program finish.
Change of intention to adhere at baseline, and at 3, 6 and 12 months after intervention. | Intervention group: measured right before and 3,6 and 12 months after the program. Control group: measured measured right before and 3,6 and 12 months after the program
  The intention to adhere is measured using a 3 items 5 points Likert scale adopted from Vissman et al. (2013). It is measured right before the interventional program begin and right after the interventional program finish.

OTHER OUTCOMES:
Qualitative evaluation on the effectiveness of the program | The selected participants will be interviewed upon 1 month after the program
  Six participants will be selected for in-depth interview. Four questions will be asked:
  1. Is the GBEP MEDIHEALTH an appropriate intervention to improve medication adherence among T2DM Malay patients? Why is it so?
  2. Does this program helped you in improving your medication adherence? If yes, how did it work?
  3. What is(are) the weakness(es) of the program and what could be done to improve it?
  4. Would you recommend this SGBI to other T2DM Malay patients?
Sustainability of the Program | Two main facilitators and the two managerial officers will be interviewed at 12 months after the program
  Two main facilitators and two managerial officers of Sarawak Pharmacy Department who are in charge of implementing the Program will be interviewed to discuss the aspects of sustainability of the Program:
  1. Manpower: Could the department sustain the manpower required in implementing the Program? How and why?
  2. Financial: Could the department sustain the long-term implementation of the Program based on the cost involved in running the Program? How and why?
  3. Organizational support: Does the aim and scope of the Program match with the long-term goals of the organisation? Does the Program gain support from top management? How and why?
  4. Reproducibility: Could the Program be easily implemented in other facilities? How and why?
  5. Demand: Is there continuous demand for the Program? How and why?

CONTACTS AND LOCATIONS:
Overall Officials: Ting Chuo Yew, MPhil, Principal Investigator — Sarawak Pharmacy Enforcement Division, Sarawak State Health Department
Locations (2):
- Malaysia (2):
  - Kota Samarahan Health Clinic, Kota Samarahan, Sarawak
  - Petra Jaya Health Clinic, Kuching, Sarawak

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers as only aggregated data will be used for the study.

REFERENCES:
- [Background] Ajzen, I. (1991). The theory of planned behavior. Organizational behavior and human decision processes, 50(2), 179-211.
- [Background] Garcia-Perez LE, Alvarez M, Dilla T, Gil-Guillen V, Orozco-Beltran D. Adherence to therapies in patients with type 2 diabetes. Diabetes Ther. 2013 Dec;4(2):175-94. doi: 10.1007/s13300-013-0034-y. Epub 2013 Aug 30. PMID 23990497
- [Background] Capoccia K, Odegard PS, Letassy N. Medication Adherence With Diabetes Medication: A Systematic Review of the Literature. Diabetes Educ. 2016 Feb;42(1):34-71. doi: 10.1177/0145721715619038. Epub 2015 Dec 4. PMID 26637240
- [Background] Meng J, Casciano R, Lee YC, Stern L, Gultyaev D, Tong L, Kitio-Dschassi B. Effect of Diabetes Treatment-Related Attributes on Costs to Type 2 Diabetes Patients in a Real-World Population. J Manag Care Spec Pharm. 2017 Apr;23(4):446-452. doi: 10.18553/jmcp.2017.23.4.446. PMID 28345434
- [Background] Alrasheedy AA, Hassali MA, Wong ZY, Saleem F. Pharmacist-managed medication therapy adherence clinics: The Malaysian experience. Res Social Adm Pharm. 2017 Jul-Aug;13(4):885-886. doi: 10.1016/j.sapharm.2017.02.011. Epub 2017 Feb 16. No abstract available. PMID 28222951
- [Background] Slater, M. D. (1999). Integrating application of media effects, persuasion, and behavior change theories to communication campaigns: A stages-of-change framework. Health Communication, 11(4), 335-354.
- [Background] Odgers-Jewell K, Ball LE, Kelly JT, Isenring EA, Reidlinger DP, Thomas R. Effectiveness of group-based self-management education for individuals with Type 2 diabetes: a systematic review with meta-analyses and meta-regression. Diabet Med. 2017 Aug;34(8):1027-1039. doi: 10.1111/dme.13340. Epub 2017 Mar 20. PMID 28226200
- [Background] Conn VS, Ruppar TM. Medication adherence outcomes of 771 intervention trials: Systematic review and meta-analysis. Prev Med. 2017 Jun;99:269-276. doi: 10.1016/j.ypmed.2017.03.008. Epub 2017 Mar 16. PMID 28315760
- [Background] Puffer S, Torgerson DJ, Watson J. Cluster randomized controlled trials. J Eval Clin Pract. 2005 Oct;11(5):479-83. doi: 10.1111/j.1365-2753.2005.00568.x. PMID 16164589
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Borek AJ, Abraham C, Smith JR, Greaves CJ, Tarrant M. A checklist to improve reporting of group-based behaviour-change interventions. BMC Public Health. 2015 Sep 25;15:963. doi: 10.1186/s12889-015-2300-6. PMID 26403082
- [Background] Fisher JD, Fisher WA, Amico KR, Harman JJ. An information-motivation-behavioral skills model of adherence to antiretroviral therapy. Health Psychol. 2006 Jul;25(4):462-73. doi: 10.1037/0278-6133.25.4.462. PMID 16846321
- [Background] Risser J, Jacobson TA, Kripalani S. Development and psychometric evaluation of the Self-efficacy for Appropriate Medication Use Scale (SEAMS) in low-literacy patients with chronic disease. J Nurs Meas. 2007;15(3):203-19. doi: 10.1891/106137407783095757. PMID 18232619
- [Derived] Ting CY, Ahmad Zaidi Adruce S, Hassali MA, Ting H, Lim CJ, Ting RS, Abd Jabar AHA, Osman NA, Shuib IS, Loo SC, Sim ST, Lim SE, Morisky DE. Effectiveness and sustainability of a structured group-based educational program (MEDIHEALTH) in improving medication adherence among Malay patients with underlying type 2 diabetes mellitus in Sarawak State of Malaysia: study protocol of a randomized controlled trial. Trials. 2018 Jun 5;19(1):310. doi: 10.1186/s13063-018-2649-9. PMID 29871651
- See also: National Use of Medicine Survey by Pharmaceutical Services Division, Ministry of Health — http://www.pharmacy.gov.my/v2/ms/dokumen/national-survey-use-medicines-nsum-malaysian-consumers-2012.html
- See also: Drug Utilization in the Treatment of Diabetes Mellitus in the Ministry of Health Facilities — http://www.pharmacy.gov.my/v2/sites/default/files/document-upload/drug-utilization-treatment-diabetes-mellitus-moh-malaysia.pdf

DOCUMENTS (1):
  • Informed Consent Form (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT03228706/ICF_002.pdf